CLINICAL TRIAL: NCT00525941
Title: An Exploratory Phase IIIb, Single-Blind, Outpatient Study to Assess Next-Day Functioning in Adult Primary Insomnia Patients Following the Administration of NBI-34060 Capsules During the Night
Brief Title: An Exploratory Study of NBI-34060 Capsules and Next Day Functioning
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to Approvable decision
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Christopher O'Brien, Chief Medical Officer, Neurocrine Biosciences, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NBI-34060-IR-0702
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NBI-34060 — 10 mg capsules; dosed as needed for falling back asleep after a bothersome awakening provided there are at least 4 hours remaining in bed; no more than one dose per night.

SUMMARY:
NBI-34060 is an investigational (research) medication being studied in people with insomnia. The current study is designed to evaluate how people, who experience a nighttime awakening with difficulty returning to sleep, feel during the next day after dosing with NBI-34060. The study will also examine the pattern and extent of nighttime awakenings as reported by the patients, as well as and the patient's sleep experience during treatment.

ELIGIBILITY:
Inclusion Criteria:

* insomnia (DSM-IV diagnosed; at least one month)
* Nocturnal awakenings
* Usual bedtimes between 9:00PM and Midnight.
* Bedtimes that do not vary by more than 2 hours on 5 or more nights per week.
* A usual time in bed of 7 to 9 hours.

Exclusion Criteria:

* no serious concomitant illness
* no other condition that could interfere with sleep

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Assessments of Next-Day Function | daily/six weeks

SECONDARY OUTCOMES:
Quality of Life | biweekly/six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Zammit, PhD, Principal Investigator — Clinilabs, Inc.
Locations (4):
- United States (4):
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Clinilabs, Inc., New York, New York
  - Community Research, Cincinnati, Ohio
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio